CLINICAL TRIAL: NCT04049201
Title: Interactive Tablet Compared to Oral Midazolam as Premedication in Preoperative Anxiety in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital d'enfants Béchir-Hamza (Other)
Responsible Party: Principal Investigator, Dr Sonia ben khalifa (PhD), clinical Professor, Hôpital d'enfants Béchir-Hamza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 02/2019
Record Dates: First submitted 2019-03-18; First posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-05

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Elective Surgical Procedures; Midazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group tablet (Experimental): group T will receive interactive Tablet containing many cartoon's videos 20 minutes before parental separation until the anesthesia induction
  Interventions: Procedure: elective surgery; Device: Interactive Tablet
- Group Midazolam (Active Comparator): group Midazolam will receive oral midazolam 0.5 mg/kg (max 20 mg) 20 minutes before the parental separation
  Interventions: Procedure: elective surgery; Drug: Midazolam

INTERVENTIONS:
Procedure: elective surgery — investigators will compare the effect of interactive tablet on preoperative anxiety in children to the effect ofMidazolam in elective surgery
  Other Names: we will study the acceptance of the facial mask,the post operative delirium and the parents satisfaction
Drug: Midazolam — Oral Midazolam
  Arms: Group Midazolam
Device: Interactive Tablet — interactive Tablet containing many cartoon's videos
  Arms: Group tablet

SUMMARY:
preoperative anxiety is an undesirable outcome in pediatric surgical patients.It can lead to behavioral trouble such as enuresis, apathy and sleep disorders.

to prevent this anxiety,many tools can be used for premedication like pharmacological:Midazolam, clonidine, hydroxysine or non pharmacological tools such as parental presence,hypnosis and interactive tablet.

the purpose of the study is to compare the effect of interactive tablet to oral midazolam.on preoperative anxiety in children prior to elective surgery

DETAILED DESCRIPTION:
this study is a prospective,randomized, active treatment controlled trial.It enrolls 100 children .

after written and informed consent,the study participants were randomly assigned using a computer generated table to one of two treatment groups prior to elective surgery.

Group T: will receive an interactive tablet containing many cartoon's videos 20 minutes before the parental separation and until the anesthesia induction Group MD:will receive oral midazolam 20 minutes before parental separation with 0.5 mg/kg (max 20mg) Anxiety assessement was done using the Modified Yale Perioperative Anxiety Scale( MYPAS) at the separation of parents,the admission in the operating room and the anesthesia induction.

Facial mask acceptance,post operative agitation (PAEDS score: Pediatric Anesthesia Emergence of Delirium) and parental satisfaction were also assessed.

ELIGIBILITY:
Inclusion Criteria:

* 3-10 years old children
* elective surgery
* ASA PS I/II

Exclusion Criteria:

* Parental refusal
* Emergency procedure
* Behavioral or psychiatric disorders
* allergy or hypersensitivity to midazolam

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2019-05-19 (Actual); Study Completion 2019-05-19 (Actual)

PRIMARY OUTCOMES:
Preoperative anxiety | 20 minutes after tablet was given
  preoperative anxiety will be measured by the modified Yale Perioperative Anxiety Scale (MYPAS)at different time prior to elective surgery .the averaged score range from 24.9: no anxiety to 100 very anxious
Preoperative anxiety | 25 minutes after tablet was given
  preoperative anxiety will be measured by the modified Yale Perioperative Anxiety Scale(MYPAS)at different time prior to elective surgery .the averaged score ranges from 24.9 no anxiety to 100 very anxious
Preoperative anxiety | 30 minutes after tablet was given
  preoperative anxiety will be measured by the modified Yale Perioperative Anxiety Scale(MYPAS)at different time prior to elective surgery.the averaged score range from 24.9 no anxiety to 100 very anxious

SECONDARY OUTCOMES:
the acceptance of Facial mask | 30 minutes after tablet was given
  the acceptance of facial mask by an established score
post operative agitation | 10 to 15 minutes after wakeup of anesthesia
  post operative agitation was assessed using PAEDS which was calculated 10 to 15 minutes after the anesthetic wake up.
the parental satisfaction | 1 hour after the wake up of anesthesia
  by an established score

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital d'Enfants Bechir Hamza, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided